CLINICAL TRIAL: NCT02861950
Title: Does Caudal Block Increase the Incidence of Urethrocutaneous Fistula Formation Following Hypospadias Repair in Infants? A Multi-center Prospective Randomized Trial.
Brief Title: Does Caudal Block Increase the Incidence of Urethrocutaneous Fistula Formation Following Hypospadias Repair in Infants?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Stanford University (Other); Dartmouth-Hitchcock Medical Center (Other); Boston Children's Hospital (Other); Children's Medical Center of Dallas/UT Southwestern (Unknown); University of Mississippi Medical Center (Other); University of New Mexico (Other); University of Michigan (Other); Children's National Research Institute (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-2343
Record Dates: First submitted 2016-06-21; First posted 2016-08-10 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Hypospadias; Urethrocutaneous Fistula
Keywords: hypospadias; caudal; urethrocutaneous fistula; penile nerve block
MeSH Terms: conditions — Hypospadias | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caudal block (Active Comparator): Patients will receive a caudal block with 0.75-1ml/kg of 0.2% ropivacaine.
  Interventions: Drug: Caudal block with ropivacaine
- Penile Nerve Block (Active Comparator): Patients will receive a dorsal penile nerve block with up to 0.75ml/kg of 0.25% bupivacaine.
  Interventions: Drug: penile nerve block with bupivacaine

INTERVENTIONS:
Drug: Caudal block with ropivacaine — Patients in this arm will receive a caudal block with ropivacaine
  Arms: Caudal block
Drug: penile nerve block with bupivacaine — Patients in this arm will receive a penile block with bupivacaine
  Arms: Penile Nerve Block

SUMMARY:
This is a prospective randomized multi-center non-inferiority trial conducted through the Pediatric Regional Anesthesia Network study sites to determine if caudal block increases the incidence of urethrocutaneous fistula following distal or mid shaft hypospadias repair compared with penile nerve block.

DETAILED DESCRIPTION:
Small retrospective series are in conflict about whether there is an association between caudal block and urethrocutaneous fistulas after hypospadias repair. The most common alternative to caudal blockade is a penile nerve block. The investigators will test the following hypothesis:

There is no difference in the incidence of urethrocutaneous fistula formation following single stage hypospadias repair with caudal anesthesia compared with penile nerve block.

The investigators will use a prospective randomized controlled design where subjects will receive either a caudal block or a penile nerve block to provide postoperative analgesia. Meatal anatomy will be graded by the urologist in the anesthetized child according to the HOPE (Hypospadias Objective Penile Evaluation) score, a validated scoring system. Both the total score and the individual component scores will be recorded. The operating urologist will determine the presence or absence of a fistula at the postoperative visit about 12 weeks after surgery, with subsequent follow up at 6 months and again at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* infants/ children with midshaft or distal hypospadias undergoing primary single stage repair in one of the Pediatric Regional Anesthesia Network participating centers.

Exclusion Criteria:

* prior hypospadias surgery,
* proximal or penoscrotal hypospadias,
* abnormal caudal anatomy or spinal dysraphism,
* cyanotic congenital heart disease,
* infection or rash at the block injection site.

Ages: 4 Months to 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of urethrocutaneous fistula | 1 year
  Presence of a urethrocutaneous fistula at postoperative visit up to 1 year after surgery.

SECONDARY OUTCOMES:
Degree of efficacy of caudal block | 1 hour after arrival in Post Anesthesia Care Unit (PACU) post surgery
  Blocks will be graded for efficacy using the following scale: Successful, Probably Successful, Probably Failed, or Failed.
Degree of pain | 1 hour after arrival in PACU post surgery
  Patients will have pain scores determined using the modified FLACC score (Face, Legs, Activity, Cry, Consolability) 1 hour after arrival in the PACU
Need for supplemental analgesics | 1 hour after arrival in PACU post surgery
  Administration of opioid in the first postoperative hour will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Megan Brockel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No